CLINICAL TRIAL: NCT02973997
Title: Combination Targeted Therapy With Pembrolizumab and Lenvatinib in Progressive, Radioiodine-Refractory Differentiated Thyroid Cancers: A Phase II Study
Brief Title: Lenvatinib and Pembrolizumab in Differentiated Thyroid Cancers (DTC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-ITOG-1504; NCI-2016-01752 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-ITOG-1504 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Results first posted 2023-10-24 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Columnar Cell Variant Thyroid Gland Papillary Carcinoma; Follicular Variant Thyroid Gland Papillary Carcinoma; Metastatic Thyroid Gland Follicular Carcinoma; Metastatic Thyroid Gland Papillary Carcinoma; Poorly Differentiated Thyroid Gland Carcinoma; Recurrent Differentiated Thyroid Gland Carcinoma; Recurrent Thyroid Gland Follicular Carcinoma; Recurrent Thyroid Gland Papillary Carcinoma; Stage III Differentiated Thyroid Gland Carcinoma AJCC v7; Stage III Thyroid Gland Follicular Carcinoma AJCC v7; Stage III Thyroid Gland Papillary Carcinoma AJCC v7; Stage IV Thyroid Gland Follicular Carcinoma AJCC v7; Stage IV Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVA Differentiated Thyroid Gland Carcinoma AJCC v7; Stage IVA Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVA Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVB Differentiated Thyroid Gland Carcinoma AJCC v7; Stage IVB Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVB Thyroid Gland Papillary Carcinoma AJCC v7; Stage IVC Differentiated Thyroid Gland Carcinoma AJCC v7; Stage IVC Thyroid Gland Follicular Carcinoma AJCC v7; Stage IVC Thyroid Gland Papillary Carcinoma AJCC v7; Tall Cell Variant Thyroid Gland Papillary Carcinoma; Thyroid Gland Hurthle Cell Carcinoma; Unresectable Differentiated Thyroid Gland Carcinoma; Unresectable Thyroid Gland Carcinoma
MeSH Terms: conditions — Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Thyroid cancer, Hurthle cell | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenvatinib, pembrolizumab) (Experimental): Patients receive lenvatinib PO QD on days 1-21 and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 19 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment for up to 35 cycles.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenvatinib; Drug: Lenvatinib Mesylate; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenvatinib — Given PO
  Other Names: E7080; ER-203492-00; Multi-Kinase Inhibitor E7080
Drug: Lenvatinib Mesylate — Given PO
  Other Names: 4-[3-Chloro-4-(N''-cyclopropylureido)phenoxy]7-methoxyquinoline-6-carboxamide Mesylate; E7080; Lenvima; Multi-Kinase Inhibitor E7080
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab and lenvatinib work in treating patients with differentiated thyroid cancer that has spread to other places in the body or has come back and cannot be removed by surgery. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the clinical efficacy, as indicated by the rate of complete response (CR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, of combination therapy with pembrolizumab and lenvatinib in lenvatinib-naive patients with progressive radioiodine-refractory differentiated thyroid cancers (DTC). (Cohort 1) II. To determine the overall response rate (ORR) by the addition of pembrolizumab to patients with radioiodine-refractory DTC who have progressive disease on lenvatinib alone. (Cohort 2)

SECONDARY OBJECTIVES:

I. To determine the safety profile and toxicity of combination therapy with pembrolizumab and lenvatinib in patients with progressive DTC. (Cohort 1 and cohort 2) II. To determine progression-free survival (PFS) and overall survival (OS). (Cohort 1 and cohort 2)

CORRELATIVE RESEARCH OBJECTIVES:

I. To correlate tumor response (RECIST 1.1) with pretreatment frequency of CD8+ T cells in the primary and/or metastatic tumor. (Cohort 1 and cohort 2) II. To correlate tumor response (RECIST 1.1) with pretreatment PD-L1 and PD-L2 levels in the primary and/or metastatic tumor. (Cohort 1 and cohort 2) III. To correlate tumor response (RECIST 1.1) with pretreatment frequency of lymphocytes expressing CD3, CD4, PD-1, FoxP3, or CD20, and of CD163+ macrophages. (Cohort 1 and cohort 2) IV. To correlate tumor response (RECIST 1.1) with the phenotype and frequency of key leukocyte subsets (i.e., PD-1+ T cells, regulatory T cells [Tregs], myeloid subsets) in the peripheral blood before, at 6 and 18 weeks on therapy, and at 54 weeks (study completion), progressive disease (PD), or study withdrawal. (Cohort 1) V. To correlate tumor response (RECIST 1.1) with PD-1+ T cell functional capacity. (Cohort 1) VI. To correlate tumor response (RECIST 1.1) with serum anti-thyroglobulin antibody levels assessed before, and at 18 weeks on therapy. (Cohort 1 and 2) VII. To correlate tumor response (RECIST 1.1) with tumor mutation status. (Cohort 1) VIII. To broadly investigate mechanisms of response and resistance to combination therapy, gene expression profiles will be generated from frozen biopsies for analysis by ribonucleic acid-sequencing (RNA-Seq). (Cohort 1)

OUTLINE:

Patients receive lenvatinib orally (PO) once daily (QD) on days 1-21 and pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 19 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment for up to 35 cycles.

After completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Locally recurrent and unresectable and/or distant metastatic differentiated thyroid cancer (DTC), histologically or cytologically confirmed; the diagnosis of DTC includes the following subtypes: papillary thyroid cancer (PTC) (including but not limited to variants such as follicular variant, tall cell, columnar cell, Hurthle cell variant of papillary carcinoma, and poorly differentiated), follicular thyroid cancer (FTC), including insular variant, Hurthle cell carcinoma and poorly differentiated thyroid cancer
* Measurable disease meeting the following criteria:

  * At least 1 lesion of >= 1.0 cm in the longest diameter for a non-lymph node or >= 1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI); if there is only one target lesion and it is a non-lymph node, it should have a longest diameter of >= 1.5 cm
  * Lesions that have had external beam radiotherapy (EBRT) or loco-regional therapies such as radiofrequency (RF) ablation must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion
* For cohort 1 only: evidence of disease progression =< 14 months prior to registration according to RECIST 1.1, as confirmed by the site study principal investigator (PI)
* For cohort 2 only: progressive disease (PD) on lenvatinib per RECIST 1.1 =< 60 days prior to registration, as confirmed by the site study PI; patients need to have documented imaging and measurement of RECIST target lesions within 30 days of starting pembrolizumab
* Radioiodine (RAI)-resistant disease as defined by one or more of the following criteria:

  * One or more measurable lesions that do not demonstrate RAI uptake
  * One or more measurable lesions progressive by RECIST 1.1 =< 14 months of prior RAI therapy
  * One or more measurable lesions present after cumulative RAI dose of >= 600 mCi
  * One or more measurable lesions that are fludeoxyglucose F-18 (FDG)-avid (> 5 standardized uptake value [SUV]), if positron emission tomography (PET)/CT scan performed; these lesions may also be RAI-avid
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count (ANC) >= 1,500 /mcL (obtained =< 30 days prior to registration)
* Platelets >= 100,000 / mcL (obtained =< 30 days prior to registration)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin dependency (=< 7 days prior to registration) (obtained =< 30 days prior to registration)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (obtained =< 30 days prior to registration)
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (obtained =< 30 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases (obtained =< 30 days prior to registration)
* Albumin >= 2.5 mg/dL (obtained =< 30 days prior to registration)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (obtained =< 30 days prior to registration)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (obtained =< 30 days prior to registration)
* Adequately controlled blood pressure with or without antihypertensive medications defined as blood pressure (BP) < 150/90 mmHg at screening
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to complete patient medication and blood pressure diaries by themselves or with assistance
* Willing and able to provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

  * Note: during the active monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Willing to provide tissue and blood samples for correlative research purposes

Exclusion Criteria:

* Cohort 1 only: prior treatment with previous VEGFR active multikinase inhibitor
* Cohort 2 only: discontinued lenvatinib due to toxicity
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Female subjects of childbearing potential: unwilling or unable to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; NOTE: subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects: unwilling or unable to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive (HIV 1/2 antibodies) and currently receiving antiretroviral therapy
* Currently participating and receiving study therapy (except lenvatinib for patients in cohort 2) or has participated in a study of an investigational agent and received study therapy within 4 weeks prior to registration
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy =< 7 days prior to the first dose of trial treatment
* Known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Prior anti-cancer monoclonal antibody (mAb) =< 4 weeks prior to registration or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered >= 4 weeks prior to registration
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 (except lenvatinib for patients in cohort 2) or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * NOTE:

    * Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
    * If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to registration, as deemed by treating investigator or site PI
* Known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis; NOTE: subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for >= 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); NOTE: replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Known history of, or any evidence of active, non-infectious pneumonitis that required steroids
* Active infection requiring systemic therapy
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Received a live vaccine =< 30 days of planned start of study therapy; NOTE: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Proteinuria > 1+ on dipstick urinalysis; patients with > 1+ proteinuria on dipstick urinalysis will undergo 24-hour urine collection for quantitative assessment; NOTE: patients with > 1 g/24 hours will be ineligible
* Clinically significant gastrointestinal malabsorption syndrome
* New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months; ejection fraction (EF) by multi-gated acquisition (MUGA) or echo should not be less than the institutional lower limit of normal
* Corrected QT (QTc) prolongation > 480 msec, as calculated by either the Bazett or Fridericia formula, as per institutional standard
* Active hemoptysis (bright red blood > 1 teaspoon on more than one occasion) =< 3 weeks prior to registration
* Cohort 2 only: more than one prior treatment with VEGFR active multikinase inhibitor prior to original start of lenvatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan R Haugen, Principal Investigator — Academic and Community Cancer Research United
Locations (7):
- United States (7):
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Baste N, Mora M, Grau JJ. Emerging systemic antitarget treatment for differentiated thyroid carcinoma. Curr Opin Oncol. 2021 May 1;33(3):184-195. doi: 10.1097/CCO.0000000000000727. PMID 33720068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two patients enrolled in cohort 2 did not begin treatment; one withdrew prior to beginning protocol treatment, and the other was found to be ineligible and was removed prior to beginning treatment.
Groups:
- Cohort 1: Lenvatinib-naïve patients
  > Patients receive lenvatinib 20mg PO QD on days 1-21 and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 19 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment for up to 35 cycles.
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Lenvatinib: Given PO
  >
  > Lenvatinib Mesylate: Given PO
  >
  > Pembrolizumab: Given IV
- Cohort 2: Previously progressed on Lenvatinib alone
  > Patients receive lenvatinib daily dose at progression QD on days 1-21 and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 19 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment for up to 35 cycles.
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Lenvatinib: Given PO
  >
  > Lenvatinib Mesylate: Given PO
  >
  > Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 30 | 25
Completed | 8 | 2
Not Completed | 22 | 23
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Adverse Event | 4 | 1
Not completed — Disease Progression | 11 | 20
Not completed — Alternative Therapy | 3 | 0
Not completed — Other complicating disease | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients were included in baseline analysis
Groups:
- Cohort 1: Lenvatinib-naïve patients> Patients receive lenvatinib 20mg PO QD on days 1-21 and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 19 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment for up to 35 cycles.> > Laboratory Biomarker Analysis: Correlative studies>
  > Lenvatinib: Given PO>
  > Lenvatinib Mesylate: Given PO>
  > Pembrolizumab: Given IV
- Cohort 2: Previously progressed on Lenvatinib alone> Patients receive lenvatinib daily dose at progression QD on days 1-21 and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 19 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment for up to 35 cycles.> > Laboratory Biomarker Analysis: Correlative studies>
  > Lenvatinib: Given PO>
  > Lenvatinib Mesylate: Given PO>
  > Pembrolizumab: Given IV
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Continuous [Median (Full Range); unit: years] | 62.5 [42 to 74] | 60 [35 to 78] | 61 [35 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 23
  Male | 14 | 20 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 24 | 21 | 45
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 30 | 27 | 57
Prior systemic VEGFR-active kinase inhibitor therapy [Count of Participants; unit: Participants]
  Yes | 0 | 24 | 24
  No | 30 | 3 | 33
Histologic subtype of primary tumor [Count of Participants; unit: Participants]
  Papillary | 19 | 11 | 30
  Follicular variant | 0 | 1 | 1
  Follicular | 3 | 1 | 4
  Hurthle | 4 | 8 | 12
  Poorly differentiated | 4 | 3 | 7
  Other | 0 | 3 | 3
ECOG Performance Status [Count of Participants; unit: Participants]
  0 - Fully active, able to carry on all pre-disease performance without restriction | 23 | 11 | 34
  1 - Restricted in strenuous activity but ambulatory and able to carry out light or sedentary work | 7 | 16 | 23

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (Cohort 1)
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Will use a one-stage binomial design.
Time Frame: 26 months
Population: All evaluable patients in cohort 1 were analyzed for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 29 | 0
percentage of participants | 0 |

2. Primary Outcome: Confirmed Response Rate (Cohort 2)
Description: Assessed by RECIST 1.1. Will use a 2-stage Simon Optimal MinMax design.
Time Frame: 27 months
Population: All evaluable patients in cohort 2 were analyzed for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 25
percentage of participants |  | 16

3. Secondary Outcome: Number of Patients Experiencing Grade 3+ Adverse Events
Description: Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03. All patients that have initiated treatment will be considered evaluable for assessing adverse events. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine adverse event patterns. Only the grade 2+ adverse events will be assessed, regardless of relationship to the study treatment.
Time Frame: 27 months
Population: All evaluable patients were analyzed for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 29 | 25
Participants | 26 | 14

4. Secondary Outcome: Progression Free Survival (PFS)
Description: The distribution of PFS will be estimated using the method of Kaplan-Meier.
Time Frame: 12 months
Population: All evaluable patients were analyzed for this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of patients alive and PF
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 29 | 25
percentage of patients alive and PF | 96.6 [90.1 to 100.0] | 48.0 [31.9 to 72.2]

5. Secondary Outcome: Overall Survival (OS)
Description: The distribution of survival at 12 months will be estimated using the method of Kaplan-Meier.
Time Frame: 12 months
Population: All evaluable patients were analyzed for this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of patients alive
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 29 | 25
percentage of patients alive | 96.6 [90.1 to 100.0] | 76.0 [61.0 to 94.7]

6. Other Pre Specified Outcome: Biomarker Levels Analysis Following Pembrolizumab and Lenvatinib Combination Therapy
Description: All analyses with respect to the translational component of this study are intended to be hypothesis-generating and descriptive in manner. Clinical data (i.e. CR rates confirmed response rates, PFS, OS, etc.) will be correlated with tumor marker data of interest (CD8+, PD-L1, PD-L2, T cell functional capacity markers, anti-thyroglobulin antibody levels, tumor mutation status, and other markers). The Chi-Square (or Fisher's Exact test) will be used to assess the association of categorical clinical data with categorical biomarker data. Time-to-event clinical data (PFS, OS) will be correlated with biomarker data using Kaplan-Meier methodology and Cox regression models. Logistic regression models will also be used to predict binary clinical data with baseline biomarker data. Finally, graphical methods and descriptive statistics will be used to summarize the data as well. Two-sided p-values < 0.05 will be considered statistically significant.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 27 months
Description: All patients that began treatment were assessed for adverse events
Groups:
- Cohort 1; Cohort 2: Pembrolizumab: Given IV
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 7/30 | 19/25
Serious Adverse Events (participants affected / at risk) | 16/30 | 8/25
Other Adverse Events (participants affected / at risk) | 30/30 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=30) | Cohort 2 (N=25)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (3)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (8) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 0 (0)
Serum amylase increased (Investigations) | 2 (2) | 0 (0)
Weight loss (Investigations) | 1 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (4) | 1 (4)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (9) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=30) | Cohort 2 (N=25)
Anemia (Blood and lymphatic system disorders) | 4 (13) | 4 (26)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (36)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (2)
Heart failure (Cardiac disorders) | 0 (0) | 1 (2)
Myocarditis (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (2)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (38) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (8) | 2 (22)
Bloating (Gastrointestinal disorders) | 1 (9) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 25 (253) | 19 (163)
Dry mouth (Gastrointestinal disorders) | 1 (18) | 1 (13)
Flatulence (Gastrointestinal disorders) | 2 (4) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (38) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 6 (10) | 1 (13)
Gingival pain (Gastrointestinal disorders) | 1 (7) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 15 (141) | 2 (15)
Nausea (Gastrointestinal disorders) | 11 (67) | 3 (58)
Oral pain (Gastrointestinal disorders) | 2 (37) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (21)
Chills (General disorders) | 2 (6) | 0 (0)
Edema face (General disorders) | 1 (9) | 0 (0)
Edema limbs (General disorders) | 2 (10) | 3 (58)
Fatigue (General disorders) | 24 (285) | 23 (302)
Fever (General disorders) | 0 (0) | 1 (6)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 9 (83) | 3 (9)
Localized edema (General disorders) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 5 (49) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (3) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 2 (4)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial throm time prolonged (Investigations) | 1 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 12 (28) | 4 (13)
Alkaline phosphatase increased (Investigations) | 4 (18) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 9 (28) | 2 (16)
Blood bilirubin increased (Investigations) | 1 (6) | 2 (7)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 6 (24) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (40) | 3 (32)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 6 (15) | 0 (0)
Weight loss (Investigations) | 22 (297) | 15 (138)
White blood cell decreased (Investigations) | 5 (9) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 18 (140) | 5 (20)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (8) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (6) | 1 (7)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (26)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (87) | 3 (60)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (15) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (13) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (6) | 2 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 8 (46) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (71) | 2 (36)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (33) | 3 (9)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (7) | 0 (0)
Dizziness (Nervous system disorders) | 1 (5) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (72) | 4 (16)
Headache (Nervous system disorders) | 8 (55) | 1 (4)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 2 (9)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (23)
Hematuria (Renal and urinary disorders) | 2 (25) | 0 (0)
Proteinuria (Renal and urinary disorders) | 11 (66) | 15 (130)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 2 (5) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (23) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (6) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 1 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 10 (141) | 1 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (27)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (14) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (14) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (31) | 1 (26)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (26) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 12 (151) | 4 (46)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (9) | 2 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (28) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 11 (78) | 3 (5)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 27 (415) | 21 (282)
Hypotension (Vascular disorders) | 2 (3) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT02973997/Prot_SAP_ICF_000.pdf